CLINICAL TRIAL: NCT01477645
Title: In Norwegian: Helseffekter av Stoff Som Avgis Ved Skyting Med HK416
Brief Title: Health Effects Following Use of Lead Free Ammunition Used With HK416
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: Norwegian Defence Research Establishment (Unknown)
Responsible Party: Principal Investigator, Svein Grahnstedt, Senior Consultant MD PhD, Oslo University Hospital
Other Study IDs: 2011/1335
Record Dates: First submitted 2011-11-18; First posted 2011-11-22 (Estimated); Last update posted 2013-10-16 (Estimated); Status verified 2013-10

CONDITIONS: Lung Function Tests; Markers of Inflammation

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Sputum and serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Leaded ammunition
- Non-leaded ammunition
- Modified non-leaded ammunition

SUMMARY:
The purpose of this study is to determine whether use of lead free ammunitions cause more respiratory problems than use of lead containing ammunitions.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers

Exclusion Criteria:

* active respiratory disease

Min Age: 20 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Voluntary army soldiers
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2011-11; Primary Completion 2012-01 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Forced Expiratory Volume (FEV1) | Before, Immediately after, and 24 hrs after exposure

SECONDARY OUTCOMES:
Inflammation markers | Before and 24 hrs after esposure

OTHER OUTCOMES:
Subjective Symptoms | During exposure, and during the 24 hrs after exposure

CONTACTS AND LOCATIONS:
Overall Officials: Kjetil Longva, PhD, Study Director — Norwegian Defence Reasearch Establishment; Anne-Katrine Borander, MD, Principal Investigator — Oslo University Hospital; Øyvind Albert Voie, PhD, Principal Investigator — Norwegian Research Defence Establishment; Johny S Kongerud, MD PhD, Study Director — Oslo University Hospital; Liv Ingunn Bjoner Sikkeland, PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Norwegian Defence Research Establishment, Kjeller, Akershus, Norway

REFERENCES:
- [Derived] Borander AK, Voie OA, Longva K, Danielsen TE, Grahnstedt S, Sandvik L, Kongerud J, Sikkeland LIB. Military small arms fire in association with acute decrements in lung function. Occup Environ Med. 2017 Sep;74(9):639-644. doi: 10.1136/oemed-2016-104207. Epub 2017 Apr 13. PMID 28408655